CLINICAL TRIAL: NCT07131449
Title: Serum Histone Succinylation as a Novel Prognostic Biomarker in Hematological Malignancies
Acronym: succinylation
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Other Study IDs: chase018; chase018 (Other: FirstAffiliatedHXinxiangMC)
Record Dates: First submitted 2025-07-15; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Leukemia; Lymphoma
Keywords: leukemia; lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient Cohort: 200 patients diagnosed with hematological malignancies: Control Cohort: 200 healthy volunteers
  Interventions: Other: This is observational studies, participants are not assigned an intervention as part of the study.

INTERVENTIONS:
Other: This is observational studies, participants are not assigned an intervention as part of the study. — This is observational studies, participants are not assigned an intervention as part of the study.

SUMMARY:
4. Study Population 4.1 Inclusion Criteria Case group

1)≥ 18 years old , regardless of gender; 2)Hematological malignancies confirmed by cytology, histology , or molecular biology , who require subsequent anti-tumor treatment ( chemotherapy , hematopoietic stem cell transplantation, radiotherapy, or cellular immunotherapy ) ; control group

1. ≥ 18 years old , regardless of gender;
2. Non-cancer patients undergoing health checkups;

4.2 Exclusion criteria

1. Pregnant women
2. Those with severe mental disorders or language communication barriers
3. Other circumstances that the researcher judges to be unsuitable for participation in this study The control group was the same as the case group V. Research Design 5.1 Overall Design This study was a single-center prospective case-control study. 5.2 Research Design Process 5.2.1 Study the specific implementation process 1. Phase 1: Screening population for enrollment i. Conduct ethical review and clinical research plan review for the project; ii. 200 patients with hematological malignancies will be selected , basic information collected , and informed consent signed ; iii: 200 healthy subjects are planned to be selected and basic information collected; 2. Second stage: Collect blood samples and perform serum histone succinylation test Blood samples were collected from all 200 eligible participants and 200 healthy subjects for serum histone succinylation testing ; 3. The third stage: statistical analysis of screening results i. Evaluate the differences in serum histone succinylation between patients with hematological malignancies and healthy controls to validate its value in early screening.

ii. Statistical analysis of the correlation between serum histone succinylation and tumor efficacy (including chemotherapy , hematopoietic stem cell transplantation, cellular immunotherapy ) and clinical outcomes . ( Efficacy evaluation was performed using RECIST 1.1 criteria )

ELIGIBILITY:
Inclusion Criteria tumor group

1. ≥ 18 years old , regardless of gender;
2. Hematological malignancies confirmed by cytology, histology , or molecular biology (such as leukemia, lymphoma, multiple myeloma, etc.), who require subsequent anti-tumor treatment ( chemotherapy , hematopoietic stem cell transplantation, radiotherapy, or cellular immunotherapy ) ; control group

1)≥ 18 years old , regardless of gender; 2)Non-cancer patients undergoing health checkups;

Exclusion criteria

1. Pregnant women
2. Those with severe mental disorders or language communication barriers
3. Other circumstances that the researcher judges to be unsuitable for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case group
  1. ≥ 18 years old , regardless of gender;
  2. Hematological malignancies confirmed by cytology, histology , or molecular biology , who require subsequent anti-tumor treatment ( chemotherapy , hematopoietic stem cell transplantation, radiotherapy, or cellular immunotherapy ) ; control group
  1)≥ 18 years old , regardless of gender; 2)Non-cancer patients undergoing health checkups;
  Exclusion criteria
  1. Pregnant women
  2. Those with severe mental disorders or language communication barriers
  3. Other circumstances that the researcher judges to be unsuitable for participation in this study The control group was the same as the case group
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the differences in serum histone succinylation levels between patients with hematologic malignancies and healthy individuals | Baseline
  To evaluate the differences in serum histone succinylation levels between patients with hematologic malignancies and healthy individuals, and to confirm whether there is a significant difference in serum histone succinylation levels between these two groups.
the correlation between serum histone succinylation modification levels and different types of tumors as well as tumor stages | through study completion, an average of 1 year
  To determine the correlation between serum histone succinylation modification levels and different types of tumors as well as tumor stages, and to statistically analyze the relationship between serum histone succinylation and therapeutic outcomes (including chemotherapy, hematopoietic stem cell transplantation, and cellular immunotherapy) as well as clinical pathological features.

CONTACTS AND LOCATIONS:
Overall Officials: guoqing LYU, Dr., Principal Investigator — The First Affiliated Hospital of Xinxiang Medical College

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-08-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT07131449/Prot_SAP_000.pdf